CLINICAL TRIAL: NCT03405467
Title: A Retrospective 10-years Nationwide Observational Study of Alpine Accidents - Flight Accidents, CPR and AED in Alpine Region, Frostbite Injuries and Lightning Strike
Brief Title: 10-years Nationwide Alpine Accidents in Austria
Status: Completed | Type: Observational
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Principal Investigator, Mathias Ströhle, Principal Investigator Dr, Medical University Innsbruck
Other Study IDs: AN4757 315/4.4
Record Dates: First submitted 2017-11-28; First posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Alpine Accident; Frostbite; Cardiopulmonary Arrest With Successful Resuscitation; Lightning Injuries; Flight Accident
MeSH Terms: conditions — Frostbite; Lightning Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- lightning accident: patients suffered injuries due to lightning strike
  Interventions: Other: general and specific data
- frostbite: patients suffered injuries due to local hypothermia leading to frostbite injuries
  Interventions: Other: general and specific data
- cpr and aed: patients suffered cardiac arrest in alpine region treated with or without automated external defibrillatior
  Interventions: Other: general and specific data
- flight accident: patients suffered injuries due to use of a flying vehicle in mountainous regions.
  Interventions: Other: general and specific data

INTERVENTIONS:
Other: general and specific data — General and specific data collected

SUMMARY:
This observational study intends to analyze the characteristic of specific accidents happened in Austrian's mountainous regions. The mechanisms of accidents which are evaluated are lightning accidents, cardiopulmonary resuscitation with or without automated external defibrillator, frostbite injuries, accidents with flying vehicle (e.g. paraglider, hang-glider…).

DETAILED DESCRIPTION:
The data are collected retrospectively from the database of Austrian alpine police force. These data are analyzed. The information from this database (scene of accident, weather, daytime…) is compared to secondary data collected from the University Hospital of Innsbruck. The comparison of both databases was approved by the Austrian Data Protection Agency. The goal of the study is to give detailed information of circumstances leading to accident and give medical information of the patient's condition and his outcome.

ELIGIBILITY:
Inclusion Criteria:

* Person suffering the injury searched for;

Exclusion Criteria:

-

Max Age: 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All Patients in the two databases eligible for the searched injury patterns.
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2015-01-21 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Number of persons suffered an accident in Alpine Mountains in Austria | 2005-2015
  The number of persons (n/year) which suffered one of the specified accidents.
Gender of persons suffered an accident in Alpine Mountains in Austria | 2005-2015
  Gender male/female or non specified which suffered one of the specified accidents.
Mortality of persons suffered an accident in Alpine Mountains in Austria | 2005-2015
  Number of persons deceased (deceased/n per year) which suffered one of the specified accidents.

SECONDARY OUTCOMES:
Number of pattern like injured patients treated in University Hospital of Innsbruck, a major tertiary trauma center in western Austria. | 2005-2015
  (n/year) treated in University Hospital of Innsbruck
Gender of pattern like injured patients treated in University Hospital of Innsbruck, a major tertiary trauma center in western Austria. | 2005-2015
  male/female, unspecified treated in University Hospital of Innsbruck
Injury severity score (ISS) of pattern like injured patients treated in University Hospital of Innsbruck, a major tertiary trauma center in western Austria. | 2005-2015
  Injury severity score of suffered injury (ISS=AIS*AIS)
Abbreviated Injury severity scale (AIS) of pattern like injured patients treated in University Hospital of Innsbruck, a major tertiary trauma center in western Austria. | 2005-2015
  Abreviated Injury severity scale of suffered injury (1-6 points; scale - minor, moderate, serious, severe, critial, maximum)
Type of evacuation and mortality | 2005-2015
  Type of evacuation (terrestrial, helicopter, combined terrestrial and helicopter) and the mortality for each group (deceased/n per year)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Paal, Dr, Principal Investigator — Hospital of Barmherzige Brüder Salzburg
Locations (1):
- General and Surgical Critical Care Medicine, Medical University of Innsbruck, Innsbruck, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Strohle M, Wallner B, Lanthaler M, Rauch S, Brugger H, Paal P. Lightning accidents in the Austrian alps - a 10-year retrospective nationwide analysis. Scand J Trauma Resusc Emerg Med. 2018 Sep 10;26(1):74. doi: 10.1186/s13049-018-0543-9. PMID 30201016